CLINICAL TRIAL: NCT05309200
Title: A Multi-Center, Randomized, Placebo-Controlled, Double-Blind, Adaptive Dose-Ranging Study to Assess Safety and Efficacy of Intravenous OCE-205 in Adults Diagnosed With Cirrhosis With Ascites Who Have Developed Hepatorenal Syndrome-Acute Kidney Injury (HRS-AKI)
Brief Title: A Study of OCE-205 in Participants With Cirrhosis With Ascites Who Developed Hepatorenal Syndrome-Acute Kidney Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocelot Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCE-205-201
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Cirrhosis; Ascites; Hepatorenal Syndrome; Acute Kidney Injury
Keywords: HRS-AKI
MeSH Terms: conditions — Fibrosis; Ascites; Hepatorenal Syndrome; Acute Kidney Injury | interventions — OCE-205

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- OCE-205 Cohort 1 (Placebo Comparator): Placebo, intravenous infusion
  Interventions: Drug: Placebo
- OCE-205 Cohort 2 (Experimental): OCE-205, 8 µg/hr, intravenous infusion
  Interventions: Drug: OCE-205
- OCE-205 Cohort 3 (Experimental): OCE-205, 15 µg/hr, intravenous infusion
  Interventions: Drug: OCE-205
- OCE-205 Cohort 4 (Experimental): OCE-205, 30 µg/hr, intravenous infusion
  Interventions: Drug: OCE-205
- OCE-205 Cohort 5 (Experimental): OCE-205, 50 µg/hr, intravenous infusion
  Interventions: Drug: OCE-205

INTERVENTIONS:
Drug: OCE-205 — The drug product, OCE-205, is a sterile solution to be used for intravenous infusion.
  Arms: OCE-205 Cohort 2; OCE-205 Cohort 3; OCE-205 Cohort 4; OCE-205 Cohort 5
Drug: Placebo — Placebo to match OCE-205 is a sterile solution to be used for intravenous infusion.
  Arms: OCE-205 Cohort 1

SUMMARY:
OCE-205 is being tested to treat participants who have developed Hepatorenal Syndrome-Acute Kidney Injury as a complication of cirrhosis with ascites.

The study aims are to evaluate the safety and efficacy of OCE-205 at various doses.

Participants will receive treatment by intravenous infusion. Participants will continue with this treatment until participants meets primary endpoint or any discontinuation criteria.

DETAILED DESCRIPTION:
The study will include 5 treatment arms including 1 Placebo Arm and 4 active drug arms. Participants will be randomly selected to 1 of 5 arms.

* Placebo
* OCE-205 at 8 micrograms per hour (µg/hr)
* OCE-205 at 15 micrograms per hour (µg/hr)
* OCE-205 at 30 micrograms per hour (µg/hr)
* OCE-205 at 50 micrograms per hour (µg/hr)

This multi-center trial will be conducted in the United States and Canada. If selected for the study, participants will be randomly assigned to 1 of the 5 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) by participant or their legal/authorized representatives.
* Diagnosed with decompensated cirrhosis with ascites.
* Receiving albumin and has had appropriate diuretic withdrawal for at least 2 days prior to randomization into the study.
* Beta-blockers should be discontinued 48 hours prior to randomization, unless doctor deems necessary for appropriate medical treatment.
* No sustained improvement in renal function after both diuretic withdrawal and plasma volume expansion with albumin.
* Female participants must have a negative pregnancy test prior to randomization and agree to avoid becoming pregnant during the study and for 30 days after the end of treatment. Male participants must agree to use 2 effective contraceptive methods during the study and up to 30 days after the end of treatment.

Exclusion Criteria:

* Serum Creatinine >3.8 mg/dL.
* Large volume paracentesis (LVP ≥6L) within 4 days of randomization.
* Pulse oximeter reading of <90% on 2L or less.
* Sepsis and/or uncontrolled bacterial infection.
* Experienced shock within 72 hrs prior to screening.
* Model for End-Stage Liver Disease (MELD) score >35.
* Hypertension with a Systolic BP > 140 mmHg and/ or a Diastolic BP >100 mmHg.
* Treated with or exposed to nephrotoxic agents or has had exposure to radiographic contrast agents within 72 hrs prior to screening.
* Has superimposed acute liver injury due to drugs, or toxins except for acute alcoholic hepatitis.
* Proteinuria greater than 500 mg/dL.
* Impaired cardiac function as evidenced by symptoms consistent with New York Heart Association Classification Class 2 or worse.
* Received Renal Replacement Therapy (RRT) within 4 weeks of randomization.
* Has had a Trans Jugular Intrahepatic Porto-systemic shunt (TIPS).
* Pregnant or breastfeeding.
* Diagnosed with a malignancy within the past 5 years.
* History or current evidence of any condition (COVID-19 positive with respiratory/cardiac complications), therapy or laboratory abnormality that might confound the results of the study, interfere with the participation for the full duration of the study, or is not in the best interest to participate in the opinion of the investigator.
* Participated in a study of an investigational medical product or device within the last 8 weeks preceding screening.
* Experienced a major blood loss (≥500 mL) within the last 4 weeks prior to screening.
* Is stuporous or comatose at screening (West Haven scores III and IV). exhibiting bradycardia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Time to measurement of concentration serum creatinine (sCr) value of less than 1.5 mg/dL on 2 consecutive days | From Day 1 infusion start to Last Day of infusion end

SECONDARY OUTCOMES:
Mean Concentration of OCE-205 at Steady State Concentration (Css) | From Day 1 infusion start to Last Day of infusion end
Rate of Total Body Clearance (CL) of OCE-205 | From Day 1 infusion start to Last Day of infusion end
Time to Elimination Half-Life (t1/2) of OCE-205 | From Day 1 infusion start to Last Day of infusion end
Volume of Steady-State Volume of Distribution (Vss) of OCE-205 | From Day 1 infusion start to Last Day of infusion end
Change in Mean Arterial Pressure (MAP) rate | From Day 1 infusion start to Last Day of infusion end
Percentage Change in rate of Mean Arterial Pressure (MAP) | From Day 1 infusion start to Last Day of infusion end
Change in Pulse Rate | From Day 1 infusion start to Last Day of infusion end
Percentage Change in Pulse Rate | From Day 1 infusion start to Last Day of infusion end
Change in concentration of Serum Creatinine (sCr) | From Day 1 infusion start to Last Day of infusion end

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Ocelot Bio
Locations (23):
- United States (22):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - Keck Medical Center of USC, Los Angeles, California
  - University of California, San Francisco Liver Clinic, San Francisco, California
  - Stanford Hospital, Stanford, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Tampa General Medical Group, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - New York-Presbyterian Hospital, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University, Dallas, Texas
  - CHI St Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angeli P, Gines P, Wong F, Bernardi M, Boyer TD, Gerbes A, Moreau R, Jalan R, Sarin SK, Piano S, Moore K, Lee SS, Durand F, Salerno F, Caraceni P, Kim WR, Arroyo V, Garcia-Tsao G. Diagnosis and management of acute kidney injury in patients with cirrhosis: revised consensus recommendations of the International Club of Ascites. J Hepatol. 2015 Apr;62(4):968-74. doi: 10.1016/j.jhep.2014.12.029. Epub 2015 Jan 28. No abstract available. PMID 25638527
- [Background] Boyer TD, Sanyal AJ, Wong F, Frederick RT, Lake JR, O'Leary JG, Ganger D, Jamil K, Pappas SC; REVERSE Study Investigators. Terlipressin Plus Albumin Is More Effective Than Albumin Alone in Improving Renal Function in Patients With Cirrhosis and Hepatorenal Syndrome Type 1. Gastroenterology. 2016 Jun;150(7):1579-1589.e2. doi: 10.1053/j.gastro.2016.02.026. Epub 2016 Feb 16. PMID 26896734
- [Background] Cavallin M, Kamath PS, Merli M, Fasolato S, Toniutto P, Salerno F, Bernardi M, Romanelli RG, Colletta C, Salinas F, Di Giacomo A, Ridola L, Fornasiere E, Caraceni P, Morando F, Piano S, Gatta A, Angeli P; Italian Association for the Study of the Liver Study Group on Hepatorenal Syndrome. Terlipressin plus albumin versus midodrine and octreotide plus albumin in the treatment of hepatorenal syndrome: A randomized trial. Hepatology. 2015 Aug;62(2):567-74. doi: 10.1002/hep.27709. Epub 2015 Feb 13. PMID 25644760
- [Background] Gines P, Sola E, Angeli P, Wong F, Nadim MK, Kamath PS. Hepatorenal syndrome. Nat Rev Dis Primers. 2018 Sep 13;4(1):23. doi: 10.1038/s41572-018-0022-7. PMID 30213943
- [Background] Martin-Llahi M, Pepin MN, Guevara M, Diaz F, Torre A, Monescillo A, Soriano G, Terra C, Fabrega E, Arroyo V, Rodes J, Gines P; TAHRS Investigators. Terlipressin and albumin vs albumin in patients with cirrhosis and hepatorenal syndrome: a randomized study. Gastroenterology. 2008 May;134(5):1352-9. doi: 10.1053/j.gastro.2008.02.024. Epub 2008 Feb 14. PMID 18471512
- [Background] McClure T, Chapman B, Hey P, Testro A, Gow P. Long-term continuous terlipressin infusion in cirrhotic patients with hepatorenal syndrome or refractory ascites awaiting liver transplantation is associated with an increase in plasma sodium. United European Gastroenterol J. 2019 Nov;7(9):1271-1273. doi: 10.1177/2050640619878996. Epub 2019 Sep 19. No abstract available. PMID 31700640
- [Background] Robertson M, Majumdar A, Garrett K, Rumler G, Gow P, Testro A. Continuous outpatient terlipressin infusion for hepatorenal syndrome as a bridge to successful liver transplantation. Hepatology. 2014 Dec;60(6):2125-6. doi: 10.1002/hep.27154. Epub 2014 May 19. No abstract available. PMID 24687396
- [Background] Salerno F, Gerbes A, Gines P, Wong F, Arroyo V. Diagnosis, prevention and treatment of hepatorenal syndrome in cirrhosis. Postgrad Med J. 2008 Dec;84(998):662-70. doi: 10.1136/gut.2006.107789. PMID 19201943
- [Background] Sanyal AJ, Boyer T, Garcia-Tsao G, Regenstein F, Rossaro L, Appenrodt B, Blei A, Gulberg V, Sigal S, Teuber P; Terlipressin Study Group. A randomized, prospective, double-blind, placebo-controlled trial of terlipressin for type 1 hepatorenal syndrome. Gastroenterology. 2008 May;134(5):1360-8. doi: 10.1053/j.gastro.2008.02.014. Epub 2008 Feb 13. PMID 18471513
- [Background] Wong F, Pappas SC, Curry MP, Reddy KR, Rubin RA, Porayko MK, Gonzalez SA, Mumtaz K, Lim N, Simonetto DA, Sharma P, Sanyal AJ, Mayo MJ, Frederick RT, Escalante S, Jamil K; CONFIRM Study Investigators. Terlipressin plus Albumin for the Treatment of Type 1 Hepatorenal Syndrome. N Engl J Med. 2021 Mar 4;384(9):818-828. doi: 10.1056/NEJMoa2008290. PMID 33657294
- [Background] Vasudevan A, Ardalan Z, Gow P, Angus P, Testro A. Efficacy of outpatient continuous terlipressin infusions for hepatorenal syndrome. Hepatology. 2016 Jul;64(1):316-8. doi: 10.1002/hep.28325. Epub 2015 Dec 22. No abstract available. PMID 26524479